CLINICAL TRIAL: NCT04209309
Title: Repetitive Transcranial Magnetic Stimulation as a Potential Tool to Reduce Sexual Arousal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Clinical Professor, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13-101-0117
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Transcranial Magnetic Stimulation
Keywords: sexual arousal
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- leDLPFC (Experimental): single session rTMS of the left dorsolateral prefrontal cortex for 15 min (60 trains with 50 stimuli; 10 sec intertrain interval; 10 Hz; 110% RMT; 3000 pulses; coil positioning over the 10-20 EEG coordinate position F3)
  Interventions: Device: repetitive transcranial magnetic stimulation
- riDLPFC (Experimental): single session rTMS of the right dorsolateral prefrontal cortex for 15 min (60 trains with 50 stimuli; 10 sec intertrain interval; 10 Hz; 110% RMT; 3000 pulses; coil positioning over the 10-20 EEG coordinate position F4)
  Interventions: Device: repetitive transcranial magnetic stimulation
- shamDLPFC (Sham Comparator): single session sham rTMS over the medial prefrontal cortex for 15 min (60 trains with 50 stimuli; 10 sec intertrain interval; 10 Hz; 110% RMT; 3000 pulses; coil positioning over the midline with tilted coil)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation

SUMMARY:
Hyper- and hyposexuality occur frequently in a variety of psychiatric disorders and are difficult to treat. While there is meta-analytic evidence for the significant effect of non-invasive brain stimulation on drug and food craving, no study has investigated the potential of this technique to modulate sexual behavior. The efficacy of a single session of high-frequency repetitive transcranial magnetic stimulation (rTMS) over the left or right dorsolateral prefrontal cortex (DLPFC) to reduce sexual arousal was tested against a sham stimulation.

To test this hypothesis, we employed a randomized, double-blind, sham-controlled crossover study design. Nineteen healthy male participants received high-frequency rTMS over the left DLPFC, high-frequency rTMS over the right DLPFC and sham rTMS (each 10 Hz; 110% resting motor threshold; 60 trains with 50 pulses) in randomized and counterbalanced order with a one-week interval between stimulation sessions to avoid carryover effects. Participants were exposed to neutral and sexual cues before and after each intervention and rated their sexual arousal after each block of cue presentation.

ELIGIBILITY:
Inclusion Criteria:

* motor threshold below 55%
* informed consent
* male
* 18-50 years
* heterosexual
* right handedness

Exclusion Criteria:

* contraindication for TMS
* somatic or mental illnesses
* intake of psychoactive drugs
* left handedness
* homo- or bisexual
* paraphilia

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change of sexual arousal | immediately before and after the single session of rTMS
  short 10-item version of the Affect and Arousal Scale, which captures perceived genital, autonomic and psychological sexual arousal as well as state sexual desire

IPD SHARING:
Plan to Share IPD: No
Not allowed based on ethics vote.